CLINICAL TRIAL: NCT00047021
Title: A Pilot Study Of Cytarabine And High-Dose Mitoxantrone For Relapsed Or Refractory Hematologic Malignancies
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent or Refractory Leukemia or Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Mary J. Laughlin, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU5Y01; P30CA043703 (NIH); CWRU-5Y01; NCI-G02-2113; CWRU-11021P; CASE-5Y01
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Leukemia; Lymphoma
Keywords: accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Recurrence; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities | interventions — sargramostim; Cytarabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: sargramostim — Sargramostim (GM-CSF) subcutaneously beginning on day 14 and continuing until blood counts recover.
Drug: cytarabine — high-dose cytarabine IV over 1 hour on days 1-5
Drug: mitoxantrone hydrochloride — high-dose mitoxantrone IV over 15-30 minutes on day 5.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining cytarabine and mitoxantrone in treating patients who have recurrent or refractory leukemia or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine non-hematologic toxic effects of high-dose cytarabine and high-dose mitoxantrone in patients with recurrent or refractory leukemia or lymphoma.
* Determine the in vitro T/NK lymphocyte proliferative responses to patient's leukemia/lymphoma cells before and after treatment with this regimen.

OUTLINE: Patients receive high-dose cytarabine IV over 1 hour on days 1-5 and high-dose mitoxantrone IV over 15-30 minutes on day 5. Patients also receive sargramostim (GM-CSF) subcutaneously beginning on day 14 and continuing until blood counts recover.

Patients who achieve at least stable disease or a response may receive a second course beginning at least 14 days after the first course is completed.

Patients are followed for 3 months.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study within approximately 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following must be present:

  * Histologically confirmed acute myeloid leukemia or acute lymphoblastic leukemia

    * More than 5% blasts in the bone marrow or peripheral blood unrelated to recovery of normal hematopoiesis from prior chemotherapy
    * Failed at least 1 attempt at induction chemotherapy
  * Diagnosis of non-Hodgkin's lymphoma or Hodgkin's lymphoma

    * Refractory or relapsed after at least 1 regimen of standard chemotherapy
  * Diagnosis of chronic myelogenous leukemia in accelerated phase or blast crisis

    * Received at least 1 myelotoxic chemotherapy regimen
* Active CNS involvement allowed

PATIENT CHARACTERISTICS:

Age

* 55 and under

Performance status

* ECOG 0-2

Life expectancy

* At least 5 weeks

Hematopoietic

* Lymphoma patients:

  * WBC at least 2,000/mm^3*
  * Platelet count at least 20,000/mm^3* NOTE: *Unless due to bone marrow involvement or disease process

Hepatic

* Bilirubin no greater than 3 times normal*
* AST/ALT no greater than 3 times normal*
* Alkaline phosphatase no greater than 3 times normal*
* No severe liver failure NOTE: *Unless related to leukemia

Renal

* Creatinine clearance greater than 50 mL/min
* No severe renal failure

Cardiovascular

* LVEF at least 45% by MUGA

Pulmonary

* DLCO at least 60% of predicted

Other

* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric illness that would preclude informed consent
* No medical illness or other condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 24 hours since prior hydroxyurea
* At least 1 week since other prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Recovered from prior therapy

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2001-11; Primary Completion 2005-08 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Event free survival at day 14 (myeloid engraftment) | day 14

SECONDARY OUTCOMES:
Incidence of serious infections by clinical, radiologic, microbiology assessment during and after treatment | followed for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary J. Laughlin, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States